CLINICAL TRIAL: NCT05041023
Title: Experience of Relatives and Caregivers of Death in ICU After the Withdrawal of Life-sustaining Therapies, Associated With an Organ Procurement Procedure (Controlled Donation After Circulatory Death).
Brief Title: Experience of Relatives and Intensive Care Units Caregivers of Controlled Donation After Circulatory Death
Acronym: CARE-M3
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence de La Biomédecine (Other Government); Fondation de France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200936
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Death, Assisted; Tissue and Organ Procurement; Life Support Care
Keywords: End-of-life; Withdrawal of life-sustaining treatments; Controlled donation after circulatory death
MeSH Terms: conditions — Suicide, Assisted; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Relative volunteers: For each situation of death of a patient in ICU following a decision to withdraw LST and for which OD has been discussed with the relatives, a relative can be included after information and acceptance of the study. One relative per situation can be included : the most involved personn in the relationship with the resuscitation team.
  Interventions: Other: Relative section
- Caregivers: For each situation of death of a patient in ICU following a decision to withdraw LST and for which OD has been considered, 2 to 3 caregivers who are present at the time the WLST is initiated can be included (1 physician and 1 or 2 paramedics).
  Interventions: Other: Caregiver section

INTERVENTIONS:
Other: Relative section — Relatives are assessed by phone calling with an experienced psychologist at 3 and 6 months after patient's death. Relatives answer to self-questionnaire and 3 scales.
  Furthermore, 20 of them are offered to participate in a semi-structured interview with an experienced psychologist, within 6 months to 1 year following the patient's death.
  Groups: Relative volunteers
Other: Caregiver section — Caregivers are self-evaluated within 72 hours after death by questionnaire survey, whose results will remain confidential to the center that included the situation.
  Furthermore, 20 of them (10 medical staff and 10 paramedical staff and / or until saturation) are offered to participate in a semi-structured interview with an experienced psychologist.
  Groups: Caregivers

SUMMARY:
Controlled donation after circulatory death (cDCD) refers to organ donation (OD) from patients whose death is defined using circulatory criteria and from whom circulatory death occurs after a planned withdrawal of life-sustaining therapies (WLST) in intensive care units (ICUs). During cDCD, the patient is still alive while OD process is being discussed and organized. Caregivers can be particularly uncomfortable in this scenario. In the specific context of cDCD, developing knowledge on the perceptions and experiences of relatives and ICU caregivers regarding OD is crucial but remains poorly investigated.

Investigators propose to conduct a prospective multicentric observational research to better understand relatives' and ICU caregivers' experience of cDCD. Better understanding their perceptions and experiences will enable to develop interventions to support and guide them throughout this practice.

DETAILED DESCRIPTION:
While withdrawal of life-sustaining therapies (WLST) decision occur significantly more frequently in intensive care units (ICUs), controlled donation after circulatory death (cDCD) evolves end-of-life care and produces a new end-of-life (EOL) model: EOL care now includes the opportunity to donate organs and tissues after death. During cDCD, the patient is still alive while OD process is being discussed and organized. Caregivers can be particularly uncomfortable in this scenario where EOL care and OD in effect overlap. Thus, the implementation of a cDCD program in France, as elsewhere, raised the issue of the potential impact of OD on WLST decision-making processes and EOL practices (particularly sedation). As other countries, the national protocol is nonetheless clear that the decision for WLST must be made in the bests interest of the patient and independent of any consideration of OD, and the donation pathway must not change EOL care. The challenge is not only to identify patients suitable as potential donors but also to provide support to grieving families and to make HCPs comfortable with OD in this particular context. In the specific context of cDCD, developing knowledge on the perceptions and experiences of relatives and ICU caregivers regarding OD is crucial but remains poorly investigated.

Investigators propose to conduct a prospective multicentric observational research to better understand relatives' and ICU caregivers' experience of cDCD.

A relative and/or at least two caregivers (1 physician and 1 or 2 paramedics) are included for any situation of death of a patient in ICU following a decision to withdraw LST and for which OD has been discussed with the relatives, whether or not the organ procurement finally occurred.

Two situations are distinguished:

* WLST without OD possibility: the WLST is initiated while OD is no longer considered for one of the following reasons: medical unsuitability, expressed intend not to be a donor or family refusal, legal issues, logistical problems, hemodynamic instability.
* WLST with OD possibility: the WLST is initiated while OD is still considered, whether or not OD finally occurs for one of the following reasons: circulatory death declared > 180 minutes, excessive warm ischemia time due to normothermic regional perfusion dysfunction or hypoperfusion.

At the time of the discussion about OD with the relatives :

* The screening for inclusion will be done.
* If 1 relative volunteers to participate in the study (non-opposition noted by the investigator), the situation is included in CARE-M3 "relative" section.
* If no relatives volunteer to participate in the study, the situation can be included in CARE M3 for the caregiver section after the patient's death.

After the patient death, wether or not OD occurs:

* 3 caregivers (1 physician and 2 paramedics) can be included. These are the caregivers who are present at the time the WLST is initiated.
* If at least two caregivers volunteer to participate in the study, the situation is included in CARE-M3 caregiver section.

Objectives concerning the relatives

* Primary objective: to study their risk of developing symptoms of post-traumatic stress disorder in the months following the patient's death.
* Secondary objectives: assessment of symptoms of anxiety, depression, complicated grief, assessment of understanding of the decision process to withdraw LST and the cDCD procedure.

Objectives concerning the ICU caregivers

* Primary objective: to study their risk developing anxiety relating to the event.
* Secondary objectives: evaluation of the impact of the cDCD procedure on the WLST decision-making process, end-of-life practices, support at the end-of-life (EOL) and quality of the EOL.

ELIGIBILITY:
Inclusion Criteria:

Any situation of anticipated death of a patient in Intensive Care Unit ICU due to circulatory arrest:

* For which a decision to withdraw Life-Sustaining Therapies LST was taken under the Claeys-Leonetti law, notified to relatives and accepted by relatives
* With a first evaluation by the hospital coordination of organ and tissue removal identifying the patient at the end of life as a potential donor: patient identified under the age of 70, with no absolute contraindication to organ removal in the context of an M3 procedure
* For which Organ Donation OD has been discussed with the relatives, whether the OD finally occurred.
* Relative and/or caregiver who has given non-objection to the use of the data.

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The relatives of patients who have died in ICU are the first attendant of the patient at the end-of-life EOL. During this procedure, relatives are particularly solicited because they are strongly involved in the decision-making process. The most involved relative in the relationship with the resuscitation team will be asked to participate in the study.
  Caregivers included in the study are caregivers from ICU who are present at the time the withdrawal of life-sustaining therapies WLST is initiated: at least 1 physician and 1 or 2 paramedics.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Hetero-evaluation of the relative using the IES-R scale | 3 months after patient's death
  Hetero-evaluation of the relative with the IES-R score (Impact of. Event Scale - Revised score). Assessment is performed by telephone interview with an experienced psychologist. This scale measures the risk for the relative of exhibiting symptoms of post-traumatic stress disorder.
Self-report of the caregiver using the STAI inventory | within 72 hours following the patient's death
  The caregiver self-assess by responding confidentially to a questionnaire: the STAI inventory (State-Trait Anxiety Inventory). This questionnaire measures their risk of developing anxiety relating to the event.

SECONDARY OUTCOMES:
Hetero-evaluation of the relative using the HADS anxiety-depression scales | 3 months after patient's death
  Hetero-evaluation of the relative with the Hospital Anxiety and Depression scales (HADS). Assessment is performed by telephone interview with an experienced psychologist. It measures symptoms of anxiety and depression.
Hetero-evaluation of the relative using the CAESAR end-of-life quality scale | 3 months after patient's death
  Hetero-evaluation of the relative with the CAESAR end-of-life quality scale which assess the quality of end-of-life care in intensive care. Assessment is performed by telephone interview with an experienced psychologist.
Hetero-evaluation of the relative using the questionnaire survey | 3 months after patient's death
  Assessment is performed by telephone interview with an experienced psychologist.
  It consists in a questionnaire of around sixty questions assessing the following themes: progress of the end-of-life process, solicitation / discussion around organ donation, understanding of the process, end-of-life experience, support, relationship with caregivers, questions a posteriori.
Hetero-evaluation of the relative using the HADS anxiety-depression scales | 6 months after patient's death
  Hetero-evaluation of the relative with the Hospital Anxiety and Depression scales (HADS). Assessment is performed by telephone interview with an experienced psychologist. It measures symptoms of anxiety and depression.
Hetero-evaluation of the relative using the IES-R scale | 6 months after patient's death
  Hetero-evaluation of the relative with the IES-R score (Impact of. Event Scale - Revised score). Assessment is performed by telephone interview with an experienced psychologist. This scale measures the risk for the relative of exhibiting symptoms of post-traumatic stress disorder.
Hetero-evaluation of the relative using the PG-13 scale | 6 months after patient's death
  Hetero-evaluation of the relative with the PG-13 scale (Prolonged Grief Disorder) which measures complicated mourning. Assessment is performed by telephone interview with an experienced psychologist.
Semi-structured interview with relative | from 6 to 12 months after patient's death
  20 relatives are selected among the included relatives to undergo a semi-structured interview conducted by an experienced psychologist in order to understand the experience of loved ones, the meaning given to the procedure, the impact of this procedure on the grieving process. These interviews will be carried out by phone call 6 months after the death within a maximum period of 12 months.
Self-evaluation of the caregiver by questionnaire survey | within 72 hours following the patient's death
  A 29-question questionnaire is completed confidentially by the caregiver. The questionnaire addresses the following topics: perception and experience of the withdrawal of life-sustaining therapies (WLST), decision-making process; perception and experience of implementing the decision; perception and experience of soliciting families; experience of the dying process; experience of the role played and involvement of different caregivers during the different stages of the process; difficulties encountered and regrets; elements of satisfaction; aspects to improve.
Semi-structured interview with caregiver | from 6 to 12 months after patient's death
  20 caregivers (10 medical staff and 10 paramedical staff and / or until saturation) are selected among the included caregivers in Ile de France to undergo a semi-structured interview conducted by an experienced psychologist.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu LE DORZE, Md, Study Director — Department of anaesthesiology and critical care medicine. Lariboisiere Hospital.
Locations (1):
- APHP - Lariboisière hospital - réanimation chirurgicale, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Dorze M, Renet A, Barthelemy R, Souppart V, Kentish-Barnes N; CARE-M3 Research Group. Relatives' experiences of end-of-life care and organ donation after controlled circulatory death: a national prospective multicenter study. Crit Care. 2025 Dec 21. doi: 10.1186/s13054-025-05807-8. Online ahead of print. PMID 41423695
- [Derived] Le Dorze M, Barthelemy R, Lesieur O, Audibert G, Azais MA, Carpentier D, Cerf C, Cheisson G, Chouquer R, Degos V, Fresco M, Lambiotte F, Mercier E, Morel J, Muller L, Parmentier-Decrucq E, Prin S, Rouhani A, Roussin F, Venhard JC, Willig M, Vernay C, Chousterman B, Kentish-Barnes N; CARE-M3 Research Group. Tensions between end-of-life care and organ donation in controlled donation after circulatory death: ICU healthcare professionals experiences. BMC Med Ethics. 2024 Oct 9;25(1):110. doi: 10.1186/s12910-024-01093-1. PMID 39385217